CLINICAL TRIAL: NCT05631249
Title: An Interventional and Translational Study Investigating Sotorasib in Previously Treated Locally Advanced or Metastatic NSCLC Subjects With Mutated KRAS p.G12C
Brief Title: Sotorasib in Previously Treated Locally Advanced or Metastatic NSCLC Subjects With Mutated KRAS p.G12C
Acronym: CODEBREAK-IGR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-006958-31; 2021/3401 (Other: CSET number); 2024-510837-16-00 (EU CTIS Number)
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: KRAS P.G12C; Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sotorasib treatment (Experimental): Sotorasib : 120 mg, once a day, per os, until progression, unacceptable toxicity, death or lost to follow-up
  Interventions: Drug: Sotorasib 120Mg Tab

INTERVENTIONS:
Drug: Sotorasib 120Mg Tab — Daily sotorasib treatment until progression, unacceptable toxicity, death, or lost to follow-up

SUMMARY:
This study aims to provide a comprehensive understanding of sotorasib's mechanisms of action and resistance in NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Age higher than 18 years;
* ECOG less or equal to 1 at the time of screening;
* Pathologically documented, previously treated, locally-advanced and unresectable or metastatic NSCLC with KRAS p.G12C mutation confirmed through molecular testing (results of both tissue and liquid biopsy are accepted);
* Subjects will have progressed or experienced disease recurrence on or after receiving at least 1 prior systemic therapy for locally advanced and unresectable or metastatic disease.
* Life expectancy of longer than 3 months from the time of screening, in the opinion of the investigator;
* Patients must have lesions easily accessible to biopsy and must have accepted to perform pre-treatment, on-treatment and end-of-treatment biopsies;
* Have adequate bone marrow reserve and organ function, based on local laboratory data within 14 days prior to registration
* Patients must understand, sign and date the written informed consent from prior to any protocol-specific procedures performed.
* Patients should be able and willing to comply with study visits and procedures as per protocol.
* Patients must be affiliated to a Social Security System or beneficiary of the same.

Exclusion Criteria:

* Patient unwilling to participate to the biological investigations and to perform biopsies and blood sample collection as required in the protocol;
* Use of known cytochrome P450 (CYP) 3A4 or P-gp sensitive substrates (with a narrow therapeutic window), within 14 days or 5 half-lives of the drug or its major active metabolite, whichever is longer, prior to registration, that was not reviewed and approved by the principal investigator.
* Use of strong inducers of CYP3A4 (including herbal supplements such as St. John's wort) within 14 days or 5 half-lives (whichever is longer) prior to registration, that was not reviewed and approved by the principal investigator.
* Inadequate washout period prior to registration, defined as: Any cytotoxic chemotherapy, investigational agents or other anticancer drug(s) from a previous cancer treatment regimen or clinical study shorter than 14 days or 5 half-lives;
* Prior treatment with a KRAS inhibitor.
* Major surgery within 28 days of registration.
* Significant gastrointestinal disorder that results in significant malabsorption, requirement for intravenous alimentation, or inability to take oral medication.
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 6 months prior to registration, unstable arrhythmias or unstable angina.
* Severe infections within 2 weeks prior to registration, but not limited to hospitalization for complications of infection, bacteremia or severe pneumonia. Prophylactic antibiotics are allowed.
* Baseline or unresolved pneumonitis from prior treatment;
* Current CTCAE version 5.0 grade higher or equal to 2 peripheral neuropathy.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures at a frequency greater than monthly. Subjects with PleurX catheters in place may be considered for the study with Principal Investigator approval.
* Known history of Human Immunodeficiency Virus (HIV) infection
* Exclusion of hepatitis infection based on the following results and/or criteria:

  1. Positive hepatitis B surface antigen (HepBsAg) (indicative of chronic Hepatitis B or recent acute hepatitis B)
  2. Negative HepBsAg with a positive for hepatitis B core antibody (Hepatitis B core antibody testing is not required for screening, however if this is done and is positive, then hepatitis B surface antibody [Anti-HBs] testing is necessary.

     Undetectable anti-HBs in this setting would suggest unclear and possible infection, and needs exclusion).
  3. Positive Hepatitis C virus antibody: Hepatitis C virus RNA by polymerase chain reaction is necessary. Detectable Hepatitis C virus RNA renders the subject ineligible.
* Leptomeningeal disease and active brain metastases. Subjects who have had brain metastases resected or have received whole brain radiation therapy or stereotactic radiosurgery ending at least 2 weeks prior to registration are eligible if they meet all of the following criteria:

  1. residual neurological symptoms grade less or equal to 2;
  2. on stable doses of dexamethasone or equivalent for at least 2 weeks, if applicable; and
  3. follow-up brain imaging performed within 30 days of enrollment shows no progression or new lesions appearing.
* Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 7 days after the last dose of sotorasib or during treatment if planning to become pregnant.
* Female subjects of childbearing potential unwilling to use 1 highly effective method of contraception during treatment and for an additional 7 days after the last dose of sotorasib
* Female subjects of childbearing potential with a positive pregnancy test assessed at Screening or day 1 by a serum pregnancy test and/or urine pregnancy test.
* Male subjects with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional 7 days after the last dose of sotorasib
* Male subjects with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for an additional 7 days after the last dose of sotorasib
* Male subjects unwilling to abstain from donating sperm during treatment and for an additional 7 days after the last dose of investigational product.
* Any evidence of primary malignancy other than locally advanced or metastatic lung cancer at within 3 years of registration, except adequately resected non-melanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated;
* Participation in another clinical trial evaluating an experimental drug (except non-interventional research).
* Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent.
* Hypersensitivity to the active substance or to any excipient
* Patients with hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2027-12-12 (Estimated); Study Completion 2027-12-12 (Estimated)

PRIMARY OUTCOMES:
Tumor response assessment | at 4 months after treatment start
  To evaluate tumor response at 4 months and decipher relevant biomarkers associated with primary (progression within the first 4 months) and acquired resistance to sotorasib (progression after 4 months).

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela ALDEA, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (5):
- France (5):
  - Centre Léon Bérard, Lyon
  - AP-HM Hôpital Nord, Marseille
  - Hôpital Paris Saint Joseph, Paris
  - AP-HP Hôpital Tenon, Paris
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No